CLINICAL TRIAL: NCT02168777
Title: A Phase 1b/2, Multi-center, Uncontrolled, Open-label, Dose Escalation Study of Refametinib (BAY86-9766) in Combination With Regorafenib (BAY73-4506) in Patients With Advanced or Metastatic Cancer
Brief Title: Refametinib (BAY86-9766) in Combination With Regorafenib (Stivarga, BAY73-4506) in Patients With Advanced or Metastatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17064; 2013-004861-15 (EudraCT Number)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2017-06

CONDITIONS: Neoplasms
Keywords: Patients with Cancer
MeSH Terms: conditions — Neoplasms | interventions — N-(3,4-difluoro-2-(2-fluoro-4-iodophenylamino)-6-methoxyphenyl)-1-(2,3-dihydroxypropyl)cyclopropane-1-sulfonamide; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ph1b-Refametinib/Regorafenib Cohort 0 (Experimental): Phase 1b part of study: Participants received different doses of Refametinib and Regorafenib combination therapy to determine recommended Phase 2 dose (RP2D) via dose-escalation. Cohort 0: Refametinib 30mg twice daily (b.i.d) + Regorafenib 80mg once daily (q.d), 3 weeks on/1 week off.
  Interventions: Drug: Refametinib (BAY86-9766); Drug: Regorafenib (Stivarga, BAY73-4506)
- Ph1b-Refametinib/Regorafenib Cohort -1 (Experimental): Phase 1b part of study: Participants received different doses of Refametinib and Regorafenib combination therapy to determine recommended Phase 2 dose (RP2D) via dose-escalation. Cohort -1: Refametinib 20mg b.i.d + Regorafenib 80mg q.d, 3 weeks on/1 week off.
  Interventions: Drug: Refametinib (BAY86-9766); Drug: Regorafenib (Stivarga, BAY73-4506)
- Ph1b-Refametinib/Regorafenib Cohort -1a (Experimental): Phase 1b part of study: Participants received different doses of Refametinib and Regorafenib combination therapy to determine recommended Phase 2 dose (RP2D) via dose-escalation. Cohort -1a: Refametinib 20mg b.i.d + Regorafenib 120mg q.d, 3 weeks on/1 week off.
  Interventions: Drug: Refametinib (BAY86-9766); Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Refametinib (BAY86-9766) — Refametinib twice daily (b.i.d.) in combination with intermittent regorafenib once daily (q.d.) at the assigned dose level.
  In Phase 2, the recommended Phase 2 dose (RP2D) for refametinib-regorafenib combination therapy will be used.
Drug: Regorafenib (Stivarga, BAY73-4506) — Refametinib twice daily (b.i.d.) in combination with intermittent regorafenib once daily (q.d.) at the assigned dose level.
  In Phase 1b dose escalation, regorafenib will be administered in a 3-weeks-on / 1-week-off schedule except in one cohort, that uses regorafenib 2 weeks on / 2 weeks off regimen (dose level -2). In Phase 2, the recommended Phase 2 dose (RP2D) for refametinib-regorafenib combination therapy will be used.

SUMMARY:
Phase I: Determine the maximum tolerated dose of combination of Regorafenib with Refametinib through a dose escalation study, all tumor types that meet certain inclusion/exclusion criteria can be entered.

After the recommended dose is determined, the Phase II portion of the study will evaluate tolerability and efficacy of the combination treatment in patients with breast cancer, lung cancer, or colorectal cancer, respectively.

DETAILED DESCRIPTION:
Number of treatment-emergent Adverse Events (AEs) will be reported in Adverse Events section.

Study was originally designed with both Phase I and Phase II part, but sponsor decided not to conduct Phase 2 part due to strategic portfolio re-prioritization.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for the Phase 1b:

  * Patients with locally advanced or metastatic solid tumors who have either relapsed following, or progressed through, standard therapy; have a current disease state for which there is no standard effective therapy; is not a candidate for, or is unwilling to undergo, standard therapy in cases where no curative option exists.
* Cohort-specific criteria for Phase 2:

  * CRC (Colorectal cancer): Patients with metastatic CRC and known KRAS (Kirsten rat sarcoma viral oncogene homolog) status who are eligible for treatment with regorafenib in accordance with the approved labeling.
  * NSCLC (Non-small-cell lung cancer): Patients with NSCLC and known KRAS status after platinum based chemotherapy.
  * Breast cancer: Patients with Her-2 negative breast cancer after anthracycline and taxane based chemotherapy.
* Baseline tumor tissue to conduct molecular and / or genetic studies should be available from all study patients enrolled in this study. (optional in Phase 1b)
* Patients must have at least one uni-dimensional measurable lesion by CT or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST)version 1.1. (applicable only in Phase 2)
* Male or female patients ≥ 18 years of age (only female patients in breast cancer cohort of Phase 2).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 3 months
* Adequate bone marrow, liver and renal function
* Cardiac function within normal range

Exclusion Criteria:

* Prior treatment with refametinib or regorafenib.
* Metastatic brain or meningeal tumors
* Uncontrolled hypertension despite optimal medical management
* History of cardiac disease
* Arterial or venous thrombotic or embolic events
* Any hemorrhage or bleeding event
* History or current evidence of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* Any condition that was unstable or which could jeopardize the safety of the patient and his/her compliance in the study.
* Excluded previous therapies and medications:

  * Radiotherapy within 3 weeks prior to start of treatment
  * Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 28 days or 5 drug half-lives (if drug half-life in patients is known), whichever is shorter (or within 6 weeks for mitomycin C) before start of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2016-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- United States (5):
  - New Haven, Connecticut
  - Detroit, Michigan
  - St Louis, Missouri
  - Chapel Hill, North Carolina
  - Houston, Texas

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was planned to have two parts, Phase 1b part and Phase 2 part. For the Phase 1b part, altogether 34 participants were screened, and 14 out of them were screening failures.
Pre-assignment Details: The remaining 20 participants were assigned to and started treatment in one of three dose escalation cohorts. The Phase 2 part was not conducted.
Period: Overall Study
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Started | 2 | 7 | 11
Completed | 0 | 0 | 0
Not Completed | 2 | 7 | 11
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Disease recurrence | 0 | 0 | 1
Not completed — Radiological disease progression | 0 | 5 | 5
Not completed — Clinical disease progression | 0 | 1 | 2
Not completed — Other reason | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a | Total
Number analyzed (Participants) | 2 | 7 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (14.1) | 56.6 (5.7) | 58.6 (7.3) | 57.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 9
  Male | 1 | 3 | 7 | 11
Cancer types [Number; unit: Participants]
  Colon and rectal cancer | 1 | 0 | 4 | 5
  Other | 1 | 2 | 2 | 5
  Non-small cell lung cancer | 0 | 3 | 1 | 4
  Breast cancer | 0 | 2 | 2 | 4
  Pancreatic adenocarcinoma | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Drug Concentration in Plasma After Multiple Dose (Cmax,md) for Refametinib
Description: Maximum drug concentration in plasma after multiple dose for Refametinib. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8 and 12 hours post-dose
Population: Pharmacokinetic (PK) analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 9
μg/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 315.9 (43) | 390.7 (52)

2. Primary Outcome: Maximum Drug Concentration in Plasma After Multiple Dose (Cmax,md) for Refametinib Metabolite M-11
Description: Maximum drug concentration in plasma after multiple dose for Refametinib metabolite M-11. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8 and 12 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 9
μg/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 104.9 (36) | 112.3 (44)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 12 h After Multiple Dose (AUC(0-12)md) for Refametinib
Description: Area under the plasma concentration-time curve from 0 to 12 h after multiple dose for Refametinib. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8 and 12 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 9
μg*h/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 2399.2 (65) | 3632.3 (51)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 12 h After Multiple Dose (AUC(0-12)md) for Refametinib Metabolite M-11
Description: Area under the plasma concentration-time curve from 0 to 12 h after multiple dose for Refametinib metabolite M-11. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8 and 12 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 9
μg*h/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 1013.4 (40) | 1144.7 (39)

5. Primary Outcome: Maximum Drug Concentration in Plasma After Multiple Dose (Cmax,md) for Regorafenib
Description: Maximum drug concentration in plasma after multiple dose for Regorafenib. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 8
μg/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 1966.0 (17) | 2206.4 (34)

6. Primary Outcome: Maximum Drug Concentration in Plasma After Multiple Dose (Cmax,md) for Regorafenib Metabolite M-2
Description: Maximum drug concentration in plasma after multiple dose for Regorafenib metabolite M-2. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 8
μg/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 1409.1 (20) | 1642.7 (98)

7. Primary Outcome: Maximum Drug Concentration in Plasma After Multiple Dose (Cmax,md) for Regorafenib Metabolite M-5
Description: Maximum drug concentration in plasma after multiple dose for Regorafenib metabolite M-5. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 8
μg/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 1148.8 (90) | 1485.7 (255)

8. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 h After Multiple Dose (AUC(0-24)md) for Regorafenib
Description: Area under the plasma concentration-time curve from 0 to 24 h after multiple dose for Regorafenib. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 8
μg*h/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 32359.4 (32) | 34352.2 (38)

9. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 h After Multiple Dose (AUC(0-24)md) for Regorafenib Metabolite M-2
Description: Area under the plasma concentration-time curve from 0 to 24 h after multiple dose for Regorafenib metabolite M-2. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 8
μg*h/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 24139.7 (34) | 25826.2 (100)

10. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 h After Multiple Dose (AUC(0-24)md) for Regorafenib Metabolite M-5
Description: Area under the plasma concentration-time curve from 0 to 24 h after multiple dose for Regorafenib metabolite M-5. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK analysis set for multiple dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 2 | 8
μg*h/L | NA (NA) — Both patients were either dose interrupted or discontinued the study. | 20531.8 (106) | 24029.3 (265)

11. Primary Outcome: Tumor Response During Phase 2 as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Tumor Response was defined as the best tumor response (Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)) observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR was defined as disappearance of tumor lesions, PR was defined as a decrease of at least 30% in the sum of tumor lesion sizes, SD was defined as steady state of disease, PD was defined as an increase of at least 20% in the sum of tumor lesions sizes.
Time Frame: Up to 12 months
Population: Phase 2 part was not conducted.
Groups:
- Ph2 - Refametinib/Regorafenib (CRC): Phase 2 part of study: Participants will receive the recommended Phase 2 dose (RP2D) for Refametinib and Regorafenib combination therapy determined in Phase 1b part. Target population for this group will be metastatic colorectal cancer (CRC).
- Ph2 - Refametinib/Regorafenib (NSCLC): Phase 2 part of study: Participants will receive the recommended Phase 2 dose (RP2D) for Refametinib and Regorafenib combination therapy determined in Phase 1b part. Target population for this group will be non-small-cell lung cancer (NSCLC).
- Ph2 - Refametinib/Regorafenib (BC): Phase 2 part of study: Participants will receive the recommended Phase 2 dose (RP2D) for Refametinib and Regorafenib combination therapy determined in Phase 1b part. Target population for this group will be Her-2 negative breast cancer (BC).
Arm/Group | Ph2 - Refametinib/Regorafenib (CRC) | Ph2 - Refametinib/Regorafenib (NSCLC) | Ph2 - Refametinib/Regorafenib (BC)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Maximum Drug Concentration in Plasma After Single (First) Dose (Cmax) for Refametinib and Its Metabolite M-11
Description: Maximum drug concentration in plasma after single (first) dose for Refametinib and its metabolite M-11. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 1 at 0 (pre-dose), 0.5, 1, 2, 4 and 8 hours post-dose
Population: PK analysis set for single dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 7 | 11
μg/L
  Refametinib | 549.7 (58) | 273.3 (82) | 253.0 (38)
  Metabolite M-11 | 58.7 (10) | 37.0 (83) | 35.7 (42)

13. Secondary Outcome: Time to Reach Maximum Drug Concentration in Plasma After Single (First) Dose (Tmax) for Refametinib and Its Metabolite M-11
Description: Time to reach maximum drug concentration in plasma after single (first) dose for Refametinib and its metabolite M-11. Median and full range were reported.
Time Frame: Cycle 1 Day 1 at 0 (pre-dose), 0.5, 1, 2, 4 and 8 hours post-dose
Population: PK analysis set for single dose.
Measure: Median (Full Range); unit: h
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 7 | 11
h
  Refametinib | 2.5 [1.00 to 4.02] | 1.0 [0.77 to 7.50] | 4.0 [0.97 to 8.00]
  Metabolite M-11 | 6.0 [4.02 to 8.00] | 4.0 [1.80 to 7.50] | 4.0 [1.93 to 8.00]

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 8 h (AUC(0-8)) After Single (First) Dose for Refametinib and Its Metabolite M-11
Description: Area under the plasma concentration-time curve from 0 to 8 h after single (first) dose for Refametinib and its metabolite M-11. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 1 at 0 (pre-dose), 0.5, 1, 2, 4 and 8 hours post-dose
Population: PK analysis set for single dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 7 | 10
μg*h/L
  Refametinib | 2377.1 (63) | 1267.9 (60) | 1314.6 (26)
  Metabolite M-11: number analyzed (Participants) | 1 | 7 | 10
  Metabolite M-11 | 411 (NA) — Summary statistic was not performed due to only one valid patient. | 212.6 (82) | 206.8 (48)

15. Secondary Outcome: Time to Reach Maximum Drug Concentration in Plasma After Multiple Dose (Tmax,md) for Refametinib and Its Metabolite M-11
Description: Time to reach maximum drug concentration in plasma after multiple dose for Refametinib and its metabolite M-11. Median and full range were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8 and 12 hours post-dose
Population: PK analysis set for multiple dose. On Day 21, one patient in Cohort 0 was dose reduced and the other patient was not dosed. Therefore no patient was evaluable.
Measure: Median (Full Range); unit: h
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 0 | 2 | 9
h
  Refametinib |  | 1.6 [1.20 to 2.00] | 4.0 [1.00 to 4.00]
  Metabolite M-11 |  | 3.0 [2.10 to 4.00] | 4.0 [0.00 to 4.03]

16. Secondary Outcome: Maximum Drug Concentration in Plasma After Single (First) Dose (Cmax) for Regorafenib and Its Metabolites M-2 and M-5
Description: Maximum drug concentration in plasma after single (first) dose for Regorafenib and its metabolites M-2 and M-5. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 1 at 0 (pre-dose), 0.5, 1, 2, 4, 8 and 24 hours post-dose
Population: PK analysis set for single dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 6 | 11
μg/L
  Regorafenib | 952.0 (34) | 794.2 (128) | 1194.6 (56)
  Metabolite M-2 | 234.4 (101) | 194.4 (438) | 367.2 (166)
  Metabolite M-5: number analyzed (Participants) | 2 | 5 | 10
  Metabolite M-5 | 22.1 (138) | 41.8 (58) | 35.1 (244)

17. Secondary Outcome: Time to Reach Maximum Drug Concentration in Plasma After Single (First) Dose (Tmax) for Regorafenib and Its Metabolites M-2 and M-5
Description: Time to reach maximum drug concentration in plasma after single (first) dose for Regorafenib and its metabolites M-2 and M-5. Median and full range were reported.
Time Frame: Cycle 1 Day 1 at 0 (pre-dose), 0.5, 1, 2, 4, 8 and 24 hours post-dose
Population: PK analysis set for single dose.
Measure: Median (Full Range); unit: h
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 6 | 11
h
  Regorafenib | 23.9 [23.75 to 23.98] | 8.0 [2.00 to 24.12] | 7.6 [2.00 to 23.95]
  Metabolite M-2 | 23.9 [23.75 to 23.98] | 8.0 [3.88 to 24.12] | 7.6 [3.97 to 25.25]
  Metabolite M-5: number analyzed (Participants) | 2 | 5 | 10
  Metabolite M-5 | 23.9 [23.75 to 23.98] | 23.6 [8.00 to 24.12] | 23.8 [23.52 to 24.17]

18. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 h (AUC(0-24)) After Single (First) Dose for Regorafenib and Its Metabolites M-2 and M-5
Description: Area under the plasma concentration-time curve from 0 to 24 h after single (first) dose for Regorafenib and its metabolites M-2 and M-5. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time Frame: Cycle 1 Day 1 at 0 (pre-dose), 0.5, 1, 2, 4, 8 and 24 hours post-dose
Population: PK analysis set for single dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/L
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 6 | 11
μg*h/L
  Regorafenib | 14642.6 (32) | 13524.8 (142) | 17475.7 (46)
  Metabolite M-2: number analyzed (Participants) | 2 | 6 | 10
  Metabolite M-2 | 3964.2 (97) | 3306.6 (452) | 6743.1 (102)
  Metabolite M-5: number analyzed (Participants) | 1 | 4 | 8
  Metabolite M-5 | 499 (NA) — Summary statistic was not performed due to only one valid patient. | 654.4 (91) | 794.2 (95)

19. Secondary Outcome: Time to Reach Maximum Drug Concentration in Plasma After Multiple Dose (Tmax,md) for Regorafenib and Its Metabolites M-2 and M-5
Description: Time to reach maximum drug concentration in plasma after multiple dose for Regorafenib and its metabolites M-2 and M-5. Median and full range were reported.
Time Frame: Cycle 1 Day 21 at 0 (pre-dose), 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 15
Measure: Median (Full Range); unit: h
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 0 | 2 | 8
h
  Regorafenib |  | 6.0 [0.00 to 12.00] | 6.0 [0.00 to 24.38]
  Metabolite M-2 |  | 11.5 [10.93 to 12.00] | 9.4 [0.00 to 24.38]
  Metabolite M-5 |  | 12.0 [0.00 to 24.08] | 9.4 [0.00 to 24.38]

20. Secondary Outcome: Tumor Response During Phase 1b as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Tumor Response was defined as the best tumor response (Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD)) observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as disappearance of all target and non-target tumor lesions, PR was defined as a decrease of at least 30% in the sum of diameters of target lesions, SD was defined neither sufficient shrinkage for PR nor sufficient increase for PD, PD was defined as an increase of at least 20% in the sum of diameters of target lesions.
Time Frame: From start of treatment until progression is documented
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 1 | 7 | 11
Participants
  Stable Disease | 1 | 2 | 5
  Progressive Disease | 0 | 5 | 6

21. Secondary Outcome: Overall Survival During Phase 2
Description: Overall survival (OS) was defined as the time (days) from the treatment start date to the date of death due to any cause. For participants who were still alive or who were lost to follow-up as of the database cutoff date for the primary completion, OS was censored at the last known alive date on or prior to the database cutoff date.
Time Frame: Up to 12 months after last patient first visit
Population: Phase 2 part was not conducted.
Arm/Group | Ph2 - Refametinib/Regorafenib (CRC) | Ph2 - Refametinib/Regorafenib (NSCLC) | Ph2 - Refametinib/Regorafenib (BC)
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Time to Progression During Phase 2
Description: Time to progression was defined as the time (days) from the treatment start date to the disease progression on or following the start date. Participants not experiencing progression at the database cutoff date for primary completion were censored at the last assessment.
Time Frame: From start of treatment until progression is documented
Population: Phase 2 part was not conducted.
Arm/Group | Ph2 - Refametinib/Regorafenib (CRC) | Ph2 - Refametinib/Regorafenib (NSCLC) | Ph2 - Refametinib/Regorafenib (BC)
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Progression-free Survival During Phase 2
Description: Progression-free survival was defined as the time from date of treatment assignment to date of first observed disease progression or death due to any cause, if death occurred while the participant was in the study and before progression was observed.
Time Frame: From start of treatment until progression is documented
Population: Phase 2 part was not conducted.
Arm/Group | Ph2 - Refametinib/Regorafenib (CRC) | Ph2 - Refametinib/Regorafenib (NSCLC) | Ph2 - Refametinib/Regorafenib (BC)
Number analyzed (Participants) | 0 | 0 | 0

24. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Dose-limiting toxicities (DLTs) were analyzed in the maximum tolerated dose (MTD) analysis set, in which only the six first patients of each dose escalation Cohort could be included according to the modified Rolling-6 method that was applied in this study.
Time Frame: At Cycle 1
Population: MTD analysis set: all participants who completed Cycle 1 or discontinued during Cycle 1 due to an adverse event or DLT in the dose escalation part.
Measure: Number; unit: Participants
Arm/Group | Ph1b-Refametinib/Regorafenib Cohort 0 | Ph1b-Refametinib/Regorafenib Cohort -1 | Ph1b-Refametinib/Regorafenib Cohort -1a
Number analyzed (Participants) | 2 | 6 | 6
Participants
  No | 0 (NA) | 6 (106) | 6 (265)
  Yes | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of study treatment until 30 days after last dose of study drug treatment.
Description: One subject had an Adverse Event which resulted in death, which was judged as unrelated to both study drugs.
Groups:
- Ph1b - Refametinib/Regorafenib Cohort 0: Phase 1b part of study: Participants received different doses of Refametinib and Regorafenib combination therapy to determine recommended Phase 2 dose (RP2D) via dose-escalation. Cohort 0: Refametinib 30mg twice daily (b.i.d) + Regorafenib 80mg once daily (q.d), 3 weeks on/1 week off.
- Ph1b - Refametinib/Regorafenib Cohort -1: Phase 1b part of study: Participants received different doses of Refametinib and Regorafenib combination therapy to determine recommended Phase 2 dose (RP2D) via dose-escalation. Cohort -1: Refametinib 20mg b.i.d + Regorafenib 80mg q.d, 3 weeks on/1 week off.
- Ph1b - Refametinib/Regorafenib Cohort -1a: Phase 1b part of study: Participants received different doses of Refametinib and Regorafenib combination therapy to determine recommended Phase 2 dose (RP2D) via dose-escalation. Cohort -1a: Refametinib 20mg b.i.d + Regorafenib 120mg q.d, 3 weeks on/1 week off.
Arm/Group | Ph1b - Refametinib/Regorafenib Cohort 0 | Ph1b - Refametinib/Regorafenib Cohort -1 | Ph1b - Refametinib/Regorafenib Cohort -1a
Serious Adverse Events (participants affected / at risk) | 0/2 | 4/7 | 5/11
Other Adverse Events (participants affected / at risk) | 2/2 | 7/7 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph1b - Refametinib/Regorafenib Cohort 0 (N=2) | Ph1b - Refametinib/Regorafenib Cohort -1 (N=7) | Ph1b - Refametinib/Regorafenib Cohort -1a (N=11)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph1b - Refametinib/Regorafenib Cohort 0 (N=2) | Ph1b - Refametinib/Regorafenib Cohort -1 (N=7) | Ph1b - Refametinib/Regorafenib Cohort -1a (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 3 (7) | 4 (7)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (3)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 3 (3) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (9) | 4 (4) | 9 (29)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 4 (8)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (3) | 2 (2) | 2 (2)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (9) | 4 (6) | 8 (24)
Malaise (General disorders) | 1 (2) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (5)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 3 (3)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Groin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastitis fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 6 (11)
Blood bilirubin increased (Investigations) | 1 (7) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (3) | 5 (12)
Blood creatinine increased (Investigations) | 0 (0) | 1 (3) | 3 (5)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 1 (1) | 1 (4) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 1 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Genital burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (2) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (8)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (3) | 3 (10)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
The sponsor decided not to conduct the Phase 2 part of the study due to strategic portfolio re-prioritization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Written consent must be obtained from Bayer prior to any information being submitted for publication. Material proposed for publication or presentation must be provided to Bayer at least 60 days prior to submission.